CLINICAL TRIAL: NCT04003142
Title: A Phase 3, Randomized, Placebo-controlled, 12-week Double-blind Study, Followed by a Non-Controlled Extension Treatment Period, to Assess the Efficacy and Safety of Fezolinetant in Women Suffering From Moderate to Severe Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Find Out if Fezolinetant Helps Reduce Moderate to Severe Hot Flashes in Women Going Through Menopause - 2
Acronym: Skylight 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-0302; 2018-003529-27 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2022-06-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Hot Flashes
Keywords: ESN364; menopause; fezolinetant; vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg (Experimental): Participants received fezolinetant 30 mg (one 30 mg fezolinetant tablet and one placebo tablet) orally, QD up to week 12 during double-blind treatment period followed by fezolinetant 30 mg orally, QD from week 13 up to Week 52 during extension treatment period.
  Interventions: Drug: Fezolinetant
- Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg (Experimental): Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD up to week 12 during double-blind treatment period followed by fezolinetant 45 mg orally, QD from week 13 up to Week 52 during extension treatment period.
  Interventions: Drug: Fezolinetant
- Double-blind Period: Placebo (Placebo Comparator): Participants received fezolinetant matching placebo (two fezolinetant matching placebo tablets) orally, once daily (QD) up to week 12 during double-blind treatment period.
  Interventions: Drug: placebo
- Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg (Experimental): Participants who received placebo during double-blind treatment period were re-randomized to receive fezolinetant 30 mg orally, QD from week 13 up to week 52 during extension treatment period.
  Interventions: Drug: Fezolinetant
- Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg (Experimental): Participants who received placebo during double-blind treatment period were re-randomized to receive fezolinetant 45 mg orally, QD from week 13 up to week 52 during extension treatment period.
  Interventions: Drug: Fezolinetant

INTERVENTIONS:
Drug: Fezolinetant — Oral tablet
  Arms: Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg; Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg; Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg; Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Drug: placebo — Oral Tablet
  Arms: Double-blind Period: Placebo

SUMMARY:
This study was for women in menopause with moderate to severe hot flashes. Menopause, a normal part of aging, is the time of a woman's last period. Hot flashes can interrupt a woman's daily life.

The study treatments are fezolinetant 30 mg (1 tablet of fezolinetant and 1 placebo tablet) once a day, fezolinetant 45 mg (2 tablets of fezolinetant) once a day or placebo (2 tablets) once a day. (Placebo is a dummy treatment that looks like medicine but does not have any medicine in it.) The study compared fezolinetant and placebo after 4 and 12 weeks of dosing. The study evaluated if fezolinetant reduces the number of hot flashes and the study evaluated if fezolinetant reduces the severity of the hot flashes.

Women in the study received an electronic handheld device at the first study visit. (It is similar to a smart phone.) Each day of the study, study participants used this to record their hot flashes. Their record for the 10 days before the start of study treatment was checked. They remained in the study if their record shows 7 or 8 moderate to severe hot flashes per day (50 or more per week). Next, they were picked for 1 of the 2 study treatments (fezolinetant or placebo) by chance alone. It is like flipping a coin.

The study participants took study treatment for 52 weeks. The first 12 weeks of study treatment was "double-blinded." That means that the study participants and the study doctors did not know who took which of the study treatments (fezolinetant 30 mg, fezolinetant 45 mg or placebo) during that time. The last 40 weeks of study treatment was "noncontrolled." That means that each study participant and the study doctors knew which study treatment that study participant took during that time. Women who took fezolinetant during the first 12 weeks continued to take the same dose. Women who took placebo during the first 12 weeks took fezolinetant. Their dose was either 30 mg or 45 mg fezolinetant.

At weeks 2, 4, 8, 12, 14, 16 and then once a month, the study participants went to the hospital or clinic for a check-up. They were asked about medications, side effects and how they felt. Other checks included physical exam and vital signs (heart rate, temperature and blood pressure). Blood and urine was collected for laboratory tests. Study participants completed questionnaires that were about how hot flashes affect their daily life. Study participants who had their uterus had the following 2 tests done at the first and last study visits. One of the 2 tests was endometrial biopsy. This test involved removing a small amount of tissue from the inside lining of the uterus. The tissue was then checked under a microscope. The other test was transvaginal ultrasound. This test used sound waves to create pictures of the organs in the pelvis. The sound waves are transmitted by a probe (transducer), which was placed inside the vagina. Study participants might have a screening mammogram done at the first and/or last study visit. A mammogram is an x-ray picture of the breasts used to screen for breast cancer. Study participants who did not have this test done in the last 12 months had it done at the first study visit. They had done at the last study visit if they were due for their screening mammogram and their own doctor agrees.

The last check-up at the hospital or clinic was 3 weeks after the last dose of study treatment.

DETAILED DESCRIPTION:
This study consisted of a screening period and a 52 week treatment period. Safety follow up occurred 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥ 18 kg/m^2 and ≤ 38 kg/m^2.
* Subject must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and confirmed as menopausal per 1 of the following criteria at the screening visit:

  * Spontaneous amenorrhea for ≥ 12 consecutive months
  * Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] > 40 IU/L); or
  * Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit.
* Within the 10 days prior to randomization, subject must have a minimum average of 7 to 8 moderate to severe hot flashes (HFs) vasomotor symptoms (VMS) per day, or 50 to 60 per week.
* Subject is in good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters, pulse rate and/or blood pressure and electrocardiogram (ECG) within the reference range for the population studied, or showing no clinically relevant deviations.
* Subject has documentation of a normal/negative or no clinically significant findings mammogram (obtained at screening or within the prior 12 months of study enrollment). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant mammographic findings.
* Subject is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and at week 52 end of treatment (EOT), and for subjects who are withdrawn from the study prior to completion, a TVU at the early discontinuation (ED) visit.
* Subject is willing to undergo an endometrial biopsy at screening and at week 52 (EOT), for subjects with uterine bleeding, and for subjects who are withdrawn from the study prior to completion. The endometrial biopsy obtained at screening must be considered evaluable.
* Subject has documentation of a normal or not clinically significant Papanicolaou (Pap) test (or equivalent cervical cytology) within the previous 12 months or at screening.
* Subject has a negative urine pregnancy test at screening.
* Subject has a negative serology panel (i.e. negative hepatitis B surface antigen, negative hepatitis C virus antibody and negative human immunodeficiency virus antibody screens) at screening.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject uses a prohibited therapy (strong or moderate cytochrome P450 1A2 [CYP1A2] inhibitors, hormone replacement therapy [HRT], hormonal contraceptive or any treatment for VMS [prescription, over the counter or herbal]) or is not willing to wash out and discontinue use of such drugs for the full duration of study conduct.
* Subject has known substance abuse or alcohol addiction within 6 months of screening.
* Subject has previous or current history of a malignant tumor, except for basal cell carcinoma.
* Subject's systolic blood pressure is ≥ 130 mmHg or diastolic blood pressure is ≥ 80 mmHg based on the average of 2 to 3 readings, on at least 2 different occasions within the screening period.

  * Subjects who do not meet these criteria may be re-assessed after initiation or review of antihypertensive measures.
  * Subjects with a medical history of hypertension can be enrolled once they are medically clear (stable and compliant).
* Subject has history of severe allergy, hypersensitivity or intolerance to drugs in general, including the study drug and any of its excipients.
* Subject has an unacceptable result from the TVU assessment at screening (i.e., full length of endometrial cavity cannot be visualized or presence of a clinically significant finding).
* Subject has an endometrial biopsy confirming presence of disordered proliferative endometrium, endometrial hyperplasia, endometrial cancer or other clinically significant findings at screening.
* Subject has a history within the last 6 months of undiagnosed uterine bleeding.
* Subject has a history of seizures or other convulsive disorders.
* Subject has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Subject has active liver disease, jaundice or elevated liver aminotransferases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total or direct bilirubin, elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP). Patients with mildly elevated ALT or AST up to 1.5 times the upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Patients with mildly elevated ALP (up to 1.5 x ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Patients with Gilbert's syndrome with elevated total bilirubin may be enrolled as long as direct bilirubin, hemoglobin and reticulocytes are normal.
* Subject has creatinine > 1.5 × ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula ≤ 59 mL/min per 1.73 m^2 at screening.
* Subject has a history of suicide attempt or suicidal behavior within the last 12 months or has suicidal ideation within the last 12 months (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale [C-SSRS]), or who is at significant risk to commit suicide at screening and at randomization.
* Subject has previously been enrolled in a clinical trial with fezolinetant.
* Subject is participating concurrently in another interventional study or participated in an interventional study within 28 days prior to screening, or received any investigational drug within 28 days or within 5 half-lives prior to screening, whichever is longer.
* Subject is unable or unwilling to complete the study procedures.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has had partial or full hysterectomy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (93):
- United States (65):
  - Mesa Obstetricians and Gynecologists, Mesa, Arizona
  - Precision Trials, Phoenix, Arizona
  - Visions Clinical Research - Tuscon, Tucson, Arizona
  - Excell Research, Oceanside, California
  - Dream Team Clinical Research, LLC, Pomona, California
  - Clinical Trials Research, Sacramento, California
  - Wake Research Associates, LLC, San Diego, California
  - Women's Healthcare Affiliates, San Diego, California
  - Bayview Research Group, Valley Village, California
  - Downtown Women's Health Care, Denver, Colorado
  - Horizons Clincial Research Center LLC, Denver, Colorado
  - Physicians' Research Options/Red Rocks OB/GYN, Lakewood, Colorado
  - Helix Biomedics, Boynton Beach, Florida
  - Renaissance Research and Medical Group, Inc., Cape Coral, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Bioclinica Research, Melbourne, Melbourne, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Suncoast Clinical Research, Inc., Miami, Florida
  - Suncoast Research, Miami, Florida
  - Medical Health Center & Research, Miami, Florida
  - Healthcare Clinical Data Inc, North Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Bioclinica Research, Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - Comprehensive Clinical Development, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Georgia Research for Women, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - WR-Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Georgia Clinical Research, Snellville, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - ASR, LLC-Advanced Specialty Research, Nampa, Idaho
  - Affinity Clinical Research Institute, Oak Brook, Illinois
  - Cypress Medical Research Center, Wichita, Kansas
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Pharmasite Research Inc, Baltimore, Maryland
  - Clinical Research Center of Nevada (CRCN), Las Vegas, Nevada
  - Dr.R. Garn Mabey, MD,Office Of, Las Vegas, Nevada
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Bosque Women's Care, Albuquerque, New Mexico
  - Circuit Clinical, West Seneca, New York
  - Premier Gynecology & Wellness, Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Hwc Women's Research Center, Englewood, Ohio
  - OB/GYN Associates of Erie, Erie, Pennsylvania
  - Dr. Marvin Kalafer MD, Office Of, Jenkintown, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - The Clinical Research Center, LLC, Carrollton, Texas
  - Advances in Health, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - FMC Science, Lampasas, Texas
  - ClinRx Research, Plano, Texas
  - Granger Medical Clinic, Riverton, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - North Spokane Women's Health, Spokane, Washington
- Canada (6):
  - Site CA15006, Sarnia, Ontario
  - Site CA15009, Toronto, Ontario
  - Site CA15007, Lévis, Quebec
  - Site CA15002, Sherbrooke, Quebec
  - Site CA15001, Victoriaville, Quebec
  - Site CA15008, Québec
- Czechia (5):
  - Site CZ42007, Písek
  - Site CZ42006, Prague
  - Site CZ42004, Prague
  - Site CZ42005, Tábor
  - Site CZ42003, Vsetín
- Latvia (2):
  - Site LV37101, Riga
  - Site LV37103, Riga
- Poland (11):
  - Site PL48001, Bydgoszcz
  - Site PL48013, Elblag
  - Site PL48009, Katowice
  - Site PL48011, Krakow
  - Site PL48002, Lublin
  - Site PL48012, Lublin
  - Site PL48004, Piaseczno
  - Site PL48006, Poznan
  - Site PL48005, Szczecin
  - Site PL48010, Warsaw
  - Site PL48003, Warsaw
- Spain (3):
  - Site ES34003, Aravaca
  - Site ES34002, Centelles
  - Site ES34001, Madrid
- Site GB44001, Shipley, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Shapiro C M M, Neal-Perry G, Stute P, Thurston RC, Wolfman W, English M, Wu X, Ottery FD. Early onset, maintenance of effect, and day-/night-time findings following fezolinetant treatment for moderate to severe vasomotor symptoms associated with menopause: A pooled phase 3 analysis. Maturitas. 2025 Dec;203:108740. doi: 10.1016/j.maturitas.2025.108740. Epub 2025 Oct 6. PMID 41259888
- [Derived] Santoro N, Neal-Perry G, Stute P, Blogg M, Mancuso S, Morga A, Ottery FD, Siddiqui E. Fezolinetant effect on vasomotor symptoms due to menopause in women unsuitable for hormone therapy. Curr Med Res Opin. 2025 Feb;41(2):375-384. doi: 10.1080/03007995.2025.2470752. Epub 2025 Mar 5. PMID 40044127
- [Derived] Kagan R, Cano A, Nappi RE, English ML, Mancuso S, Wu X, Ottery FD. Safety of Fezolinetant for Treatment of Moderate to Severe Vasomotor Symptoms Due to Menopause: Pooled Analysis of Three Randomized Phase 3 Studies. Adv Ther. 2025 Feb;42(2):1147-1164. doi: 10.1007/s12325-024-03073-8. Epub 2024 Dec 30. PMID 39739195
- [Derived] Morga A, Zimmermann L, Valluri U, Siddiqui E, McLeod L, Bender RH. Validation and Application of Thresholds to Define Meaningful Change in Vasomotor Symptoms Frequency: Analysis of Pooled SKYLIGHT 1 and 2 Data. Adv Ther. 2024 Jul;41(7):2845-2858. doi: 10.1007/s12325-024-02849-2. Epub 2024 May 22. PMID 38775925
- [Derived] Schultz NM, Morga A, Siddiqui E, Rhoten SE. Psychometric Evaluation of the MENQOL Instrument in Women Experiencing Vasomotor Symptoms Associated with Menopause. Adv Ther. 2024 Jun;41(6):2233-2252. doi: 10.1007/s12325-024-02787-z. Epub 2024 Feb 24. PMID 38396203
- [Derived] Schultz NM, Morga A, Siddiqui E, Rhoten SE. Psychometric evaluation of the PROMIS SD-SF-8b instrument in individuals experiencing vasomotor symptoms due to menopause. Health Qual Life Outcomes. 2023 Nov 21;21(1):126. doi: 10.1186/s12955-023-02206-x. PMID 37990323
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14833&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women participants 40 to 65 years of age who had moderate to severe vasomotor symptoms (VMS) and seeking treatment or relief for VMS associated with menopause, confirmed as menopausal, had to have 7 to 8 moderate to severe VMS per day within the 10 days prior to randomization and who met the inclusion criteria and none of the exclusion criteria were enrolled in this study.
Pre-assignment Details: Prior to randomization, participants had a screening period during which a minimum 10-day collection of baseline VMS frequency and severity assessments were performed.
Period: Double-blind Period (12 Weeks)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Started | 168 | 166 | 167 | 0 | 0
Treated | 167 | 166 | 167 | 0 | 0
Completed | 151 | 152 | 155 | 0 | 0
Not Completed | 17 | 14 | 12 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0 | 0
Not completed — Protocol Deviation | 1 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 6 | 6 | 0 | 0
Not completed — Miscellaneous | 2 | 1 | 2 | 0 | 0
Period: Extension Period (40 Weeks)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Started | 0 (Participants who received placebo in double-blind period were moved to fezolinetant 30/45 mg arms in extension treatment period) | 152 | 154 (One participant who completed double-blind period discontinued the study before entering the extension treatment period.) | 76 (Participants who received placebo in double-blind period were randomized to fezolinetant 30 mg arms) | 75 (Participants who received placebo in double-blind period were randomized to fezolinetant 45 mg arms)
Completed | 0 | 125 | 132 | 63 | 63
Not Completed | 0 | 27 | 22 | 13 | 12
Not completed — Adverse Event | 0 | 4 | 4 | 2 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 2 | 1
Not completed — Protocol Deviation | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 17 | 14 | 9 | 5
Not completed — Miscellaneous | 0 | 4 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg: Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD up to week 12 during double-blind treatment period followed by fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD from week 13 up to Week 52 during extension treatment period.
- Total: Total of all reporting groups
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Total
Number analyzed (Participants) | 168 | 166 | 167 | 501
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (4.6) | 53.9 (4.9) | 54.3 (5.4) | 54.3 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 166 | 167 | 501
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 34 | 41 | 108
  Not Hispanic or Latino | 134 | 132 | 126 | 392
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 31 | 35 | 33 | 99
  White | 135 | 131 | 132 | 398
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Frequency of Moderate and Severe VMS per 24 hours [Mean (Standard Deviation); unit: VMS per day] — The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Population: Full analysis set (FAS) consisted of all randomized participants who took at least 1 dose of study intervention.
  VMS per day
    number analyzed (Participants) | 167 | 166 | 167 | 500
    (all) | 11.59 (5.02) | 11.23 (4.88) | 11.79 (8.26) | 11.54 (6.25)
Severity of Moderate and Severe VMS per 24 hours [Mean (Standard Deviation); unit: Score on a scale] — Severity of moderate to severe VMS per day was calculated as follows: [(number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily moderate/severe VMS. Higher score indicates greater severity. Baseline was the weighted average of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization Population: FAS population
  Score on a scale
    number analyzed (Participants) | 167 | 166 | 167 | 500
    (all) | 2.41 (0.32) | 2.44 (0.33) | 2.41 (0.34) | 2.42 (0.33)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in The Mean Frequency of Moderate to Severe VMS at Week 4
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization.
Time Frame: Baseline and week 4
Population: Full analysis set (FAS) (consisted of all randomized participants who took at least 1 dose of study intervention) with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Groups:
- Double-blind Period: Fezolinetant 30 mg: Participants received fezolinetant 30 mg (one 30 mg fezolinetant tablet and one placebo tablet) orally, QD up to week 12 during double-blind treatment.
- Double-blind Period: Fezolinetant 45 mg: Participants received fezolinetant 45 mg (one 30 mg tablet and one 15 mg tablet) orally, QD up to week 12 during double-blind treatment period.
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 151 | 155 | 155
VMS per day | -3.72 (0.33) | -5.53 (0.33) | -6.26 (0.33)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority — Least squares Mean (LSM), Standard error (SE), Confidence interval (CI), Mixed model repeated measures (MMRM), Change from Baseline (CFB), Dependent variable (dv), Treatment (tr), Week (wk), Baseline (bl), Weight (wt); p < 0.001, MMRM — LSM, SE, CI, & p-values come from MMRM analysis of covariance model with CFB as dv & trt group, wk & smoking status as factors, with bl measurement & bl wt as covariates, as well as an interaction of trt by wk & interaction of bl measurement by wk; Least squares (LS) Mean difference = -1.82, 95% CI 2-sided [-2.73 to -0.91], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.55, 95% CI [-3.45 to -1.64], Standard Error of Mean 0.46
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.049, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, Hochberg

2. Primary Outcome: Change From Baseline in The Mean Frequency of Moderate to Severe VMS at Week 12
Description: as for outcome 1
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 140 | 133 | 145
VMS per day | -4.97 (0.39) | -6.83 (0.39) | -7.50 (0.39)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean Difference = -1.86, 95% CI [-2.94 to -0.78], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.53, 95% CI 2-sided [-3.60 to -1.46], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.049, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, Hochberg

3. Primary Outcome: Change From Baseline in The Mean Severity of Moderate to Severe VMS at Week 4
Description: Severity of moderate to severe VMS per day at post baseline visit was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]/Total number of daily mild/moderate/severe hot flashes Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
  Severity was zero for participants that had no mild or moderate or severe VMS. Higher scores indicates greater severity.
Time Frame: Baseline and week 4
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 151 | 155 | 155
Score on a scale | -0.32 (0.05) | -0.47 (0.05) | -0.61 (0.05)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.021, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.15, 95% CI [-0.27 to -0.02], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.29, 95% CI [-0.41 to -0.16], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.049, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, Hochberg

4. Primary Outcome: Change From Baseline in The Mean Severity of Moderate to Severe VMS at Week 12
Description: as for outcome 3
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 140 | 133 | 145
Score on a scale | -0.48 (0.06) | -0.64 (0.06) | -0.77 (0.06)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.049, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.16, 95% CI [-0.33 to 0.00], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.29, 95% CI [-0.45 to -0.13], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.049, Hochberg
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p < 0.001, Hochberg

5. Secondary Outcome: Change From Baseline in The Mean Patient-reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b) Total Score at Week 12
Description: The PROMIS SD SF 8b assesses self-reported sleep disturbance over the past 7 days and includes perceptions of restless sleep; satisfaction with sleep; refreshing sleep; difficulties sleeping, getting to sleep or staying asleep; amount of sleep; and sleep quality. Because it assesses the participants experience of sleep disturbance, the measure does not focus on specific sleep-disorder symptoms or ask participants to report objective measures of sleep (e.g., total amount of sleep, time to fall asleep and amount of wakefulness during sleep). Responses to each of the 8 items range from 1 (no disturbed sleep) to 5 (disturbed sleep), and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS SD SF 8b indicate more of the disturbed sleep.
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 143 | 139 | 145
Score on a scale | -3.4 (0.5) | -4.1 (0.5) | -5.5 (0.5)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Test type: Superiority; p = 0.381, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-2.1 to 0.8], Standard Error of Mean 0.7
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.5 to -0.6], Standard Error of Mean 0.7

6. Secondary Outcome: Change From Baseline in The Mean Frequency of Moderate, and Severe VMS to Each Study Week Up to Week 12
Description: as for outcome 1
Time Frame: Baseline and weeks 1, 2, 3, 5, 6, 7, 8, 9, 10, and 11
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 166 | 164 | 158
VMS per day
  Week 1 | -2.32 (0.28) | -3.62 (0.29) | -4.03 (0.29)
  Week 2: number analyzed (Participants) | 159 | 160 | 156
  Week 2 | -3.06 (0.32) | -4.82 (0.32) | -5.03 (0.32)
  Week 3: number analyzed (Participants) | 156 | 157 | 156
  Week 3 | -3.56 (0.32) | -5.29 (0.32) | -5.95 (0.32)
  Week 5: number analyzed (Participants) | 152 | 152 | 154
  Week 5 | -4.05 (0.34) | -5.89 (0.34) | -6.71 (0.34)
  Week 6: number analyzed (Participants) | 152 | 146 | 149
  Week 6 | -4.25 (0.33) | -6.03 (0.33) | -6.91 (0.33)
  Week 7: number analyzed (Participants) | 149 | 143 | 147
  Week 7 | -4.44 (0.35) | -6.24 (0.35) | -6.78 (0.35)
  Week 8: number analyzed (Participants) | 148 | 143 | 154
  Week 8 | -4.48 (0.37) | -6.25 (0.37) | -6.86 (0.37)
  Week 9: number analyzed (Participants) | 145 | 140 | 148
  Week 9 | -4.88 (0.38) | -6.54 (0.38) | -7.39 (0.38)
  Week 10: number analyzed (Participants) | 139 | 138 | 149
  Week 10 | -4.83 (0.38) | -6.74 (0.38) | -7.47 (0.38)
  Week 11: number analyzed (Participants) | 138 | 142 | 149
  Week 11 | -4.90 (0.38) | -6.76 (0.38) | -7.46 (0.37)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.30, 95% CI 2-sided [-2.09 to -0.51], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.71, 95% CI [-2.51 to -0.91], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.76, 95% CI [-2.65 to -0.87], Standard Error of Mean 0.45
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.97, 95% CI [-2.86 to -1.08], Standard Error of Mean 0.45
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.74, 95% CI [-2.63 to -0.84], Standard Error of Mean 0.46
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.40, 95% CI [-3.29 to -1.50], Standard Error of Mean 0.46
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.84, 95% CI [-2.79 to -0.90], Standard Error of Mean 0.48
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.66, 95% CI 2-sided [-3.61 to -1.72], Standard Error of Mean 0.48
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.78, 95% CI 2-sided [-2.71 to -0.85], Standard Error of Mean 0.47
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.66, 95% CI [-3.59 to -1.73], Standard Error of Mean 0.47
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.80, 95% CI [-2.77 to -0.83], Standard Error of Mean 0.49
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.34, 95% CI [-3.30 to -1.37], Standard Error of Mean 0.49
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.76, 95% CI 2-sided [-2.79 to -0.74], Standard Error of Mean 0.52
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.38, 95% CI 2-sided [-3.40 to -1.35], Standard Error of Mean 0.52
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.65, 95% CI [-2.71 to -0.59], Standard Error of Mean 0.54
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.51, 95% CI [-3.57 to -1.45], Standard Error of Mean 0.54
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.91, 95% CI [-2.96 to -0.86], Standard Error of Mean 0.54
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.65, 95% CI [-3.69 to -1.60], Standard Error of Mean 0.53
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.86, 95% CI [-2.91 to -0.81], Standard Error of Mean 0.53
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -2.56, 95% CI 2-sided [-3.61 to -1.52], Standard Error of Mean 0.53

7. Secondary Outcome: Change From Baseline in The Mean Severity of Moderate, and Severe VMS to Each Study Week Up to Week 12
Description: as for outcome 3
Time Frame: Baseline and weeks 1, 2, 3, 5, 6, 7, 8, 9, 10 and 11
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 166 | 164 | 158
Score on a scale
  Week 1 | -0.18 (0.03) | -0.32 (0.03) | -0.34 (0.03)
  Week 2: number analyzed (Participants) | 159 | 160 | 156
  Week 2 | -0.24 (0.04) | -0.41 (0.04) | -0.42 (0.04)
  Week 3: number analyzed (Participants) | 156 | 157 | 156
  Week 3 | -0.31 (0.04) | -0.42 (0.04) | -0.54 (0.04)
  Week 5: number analyzed (Participants) | 152 | 152 | 154
  Week 5 | -0.37 (0.05) | -0.53 (0.05) | -0.66 (0.05)
  Week 6: number analyzed (Participants) | 152 | 146 | 149
  Week 6 | -0.37 (0.05) | -0.55 (0.05) | -0.65 (0.05)
  Week 7: number analyzed (Participants) | 149 | 143 | 147
  Week 7 | -0.42 (0.05) | -0.58 (0.05) | -0.70 (0.05)
  Week 8: number analyzed (Participants) | 148 | 143 | 154
  Week 8 | -0.43 (0.05) | -0.56 (0.05) | -0.69 (0.05)
  Week 9: number analyzed (Participants) | 145 | 140 | 148
  Week 9 | -0.46 (0.06) | -0.59 (0.06) | -0.74 (0.06)
  Week 10: number analyzed (Participants) | 139 | 138 | 149
  Week 10 | -0.45 (0.06) | -0.64 (0.06) | -0.76 (0.06)
  Week 11: number analyzed (Participants) | 138 | 142 | 149
  Week 11 | -0.46 (0.06) | -0.67 (0.06) | -0.77 (0.06)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.13, 95% CI [-0.21 to -0.05], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.16, 95% CI 2-sided [-0.24 to -0.08], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.17, 95% CI [-0.28 to -0.07], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.18, 95% CI 2-sided [-0.28 to -0.07], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p = 0.067, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.11, 95% CI [-0.23 to 0.01], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.23, 95% CI 2-sided [-0.35 to -0.11], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p = 0.020, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.16, 95% CI 2-sided [-0.30 to -0.03], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.29, 95% CI 2-sided [-0.43 to -0.16], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p = 0.012, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.18, 95% CI 2-sided [-0.32 to -0.04], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.28, 95% CI [-0.42 to -0.14], Standard Error of Mean 0.07
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p = 0.030, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.16, 95% CI 2-sided [-0.31 to -0.02], Standard Error of Mean 0.07
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.28, 95% CI 2-sided [-0.43 to -0.14], Standard Error of Mean 0.07
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p = 0.095, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.13, 95% CI 2-sided [-0.28 to 0.02], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.26, 95% CI 2-sided [-0.41 to -0.11], Standard Error of Mean 0.08
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.109, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.13, 95% CI 2-sided [-0.28 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.28, 95% CI 2-sided [-0.43 to -0.12], Standard Error of Mean 0.08
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p = 0.020, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.19, 95% CI [-0.35 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.31, 95% CI [-0.47 to -0.15], Standard Error of Mean 0.08
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p = 0.012, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean diferrence = -0.21, 95% CI [-0.37 to -0.05], Standard Error of Mean 0.08
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.31, 95% CI [-0.47 to -0.15], Standard Error of Mean 0.08

8. Secondary Outcome: Mean Percent Change in The Frequency of Moderate And Severe Vasomotor Symptoms From Baseline to Each Study Week Up to Week 12
Description: as for outcome 1
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 166 | 164 | 158
Percent change
  Week 1 | -20.82 (2.42) | -32.98 (2.43) | -36.50 (2.45)
  Week 2: number analyzed (Participants) | 159 | 160 | 156
  Week 2 | -29.21 (2.69) | -43.82 (2.69) | -45.16 (2.71)
  Week 3: number analyzed (Participants) | 156 | 157 | 156
  Week 3 | -33.17 (2.76) | -48.68 (2.75) | -53.42 (2.76)
  Week 4: number analyzed (Participants) | 151 | 155 | 155
  Week 4 | -34.72 (2.78) | -51.06 (2.77) | -56.37 (2.77)
  Week 5: number analyzed (Participants) | 152 | 152 | 154
  Week 5 | -37.88 (2.75) | -53.50 (2.75) | -60.76 (2.74)
  Week 6: number analyzed (Participants) | 152 | 146 | 149
  Week 6 | -39.64 (2.73) | -54.42 (2.73) | -62.30 (2.73)
  Week 7: number analyzed (Participants) | 149 | 143 | 147
  Week 7 | -40.91 (2.84) | -55.88 (2.84) | -62.38 (2.83)
  Week 8: number analyzed (Participants) | 148 | 143 | 154
  Week 8 | -41.84 (2.86) | -56.22 (2.86) | -62.42 (2.84)
  Week 9: number analyzed (Participants) | 145 | 140 | 148
  Week 9 | -45.87 (2.88) | -58.01 (2.88) | -65.60 (2.86)
  Week 10: number analyzed (Participants) | 139 | 138 | 149
  Week 10 | -45.58 (2.83) | -59.98 (2.82) | -65.68 (2.81)
  Week 11: number analyzed (Participants) | 138 | 142 | 149
  Week 11 | -45.41 (2.88) | -60.37 (2.87) | -65.56 (2.86)
  Week 12: number analyzed (Participants) | 140 | 133 | 145
  Week 12 | -46.91 (2.87) | -60.55 (2.87) | -65.85 (2.85)
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -12.16, 95% CI [-18.90 to -5.43], Standard Error of Mean 3.43
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -15.68, 95% CI [-22.44 to -8.91], Standard Error of Mean 3.44
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -14.61, 95% CI 2-sided [-22.09 to -7.13], Standard Error of Mean 3.81
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -15.95, 95% CI 2-sided [-23.45 to -8.45], Standard Error of Mean 3.82
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -15.51, 95% CI [-23.16 to -7.86], Standard Error of Mean 3.89
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -20.25, 95% CI [-27.91 to -12.59], Standard Error of Mean 3.90
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 4; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -16.34, 95% CI [-24.04 to -8.63], Standard Error of Mean 3.92
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 4; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -21.65, 95% CI [-29.36 to -13.94], Standard Error of Mean 3.92
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -15.62, 95% CI 2-sided [-23.27 to -7.98], Standard Error of Mean 3.89
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -22.88, 95% CI [-30.52 to -15.24], Standard Error of Mean 3.89
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -14.78, 95% CI [-22.38 to -7.19], Standard Error of Mean 3.87
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -22.66, 95% CI 2-sided [-30.25 to -15.07], Standard Error of Mean 3.86
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -14.97, 95% CI 2-sided [-22.86 to -7.09], Standard Error of Mean 4.01
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -21.47, 95% CI [-29.34 to -13.60], Standard Error of Mean 4.01
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -14.38, 95% CI 2-sided [-22.33 to -6.43], Standard Error of Mean 4.05
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -20.57, 95% CI [-28.50 to -12.65], Standard Error of Mean 4.03
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -12.14, 95% CI [-20.14 to -4.14], Standard Error of Mean 4.07
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -19.73, 95% CI 2-sided [-27.71 to -11.755], Standard Error of Mean 4.06
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -14.40, 95% CI 2-sided [-22.25 to -6.54], Standard Error of Mean 4.0
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -20.10, 95% CI [-27.93 to -12.27], Standard Error of Mean 3.98
Statistical Analysis 21: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -14.96, 95% CI [-22.96 to -6.96], Standard Error of Mean 4.07
Statistical Analysis 22: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -20.15, 95% CI 2-sided [-28.13 to -12.18], Standard Error of Mean 4.06
Statistical Analysis 23: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 12; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -13.64, 95% CI [-21.62 to -5.65], Standard Error of Mean 4.07
Statistical Analysis 24: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 12; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -18.94, 95% CI [-26.89 to -10.98], Standard Error of Mean 4.05

9. Secondary Outcome: Number of Participants With Percent Reduction of >=50% in the Mean Frequency of Moderate and Severe VMS From Baseline to Each Study Week Up to Week 12
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Participant has >=50% reduction from baseline to each post baseline week for the frequency of moderate to severe VMS.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 167 | 166 | 167
Participants
  Week 1 | 28 | 46 | 58
  Week 2 | 39 | 71 | 71
  Week 3 | 48 | 81 | 89
  Week 4 | 44 | 84 | 88
  Week 5 | 54 | 84 | 98
  Week 6 | 53 | 81 | 95
  Week 7 | 55 | 84 | 92
  Week 8 | 56 | 81 | 103
  Week 9 | 64 | 84 | 98
  Week 10 | 62 | 85 | 103
  Week 11 | 60 | 94 | 105
  Week 12 | 71 | 84 | 101
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p = 0.020, Regression, Logistic — Based on logistic regression with treatment group and smoking status (current vs former/never) as factors and mean frequency of vasomotor symptoms at baseline as a covariate; Odds Ratio (OR) = 1.881, 95% CI [1.110 to 3.233]
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.645, 95% CI 2-sided [1.585 to 4.498]
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.464, 95% CI [1.535 to 4.001]
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.464, 95% CI 2-sided [1.534 to 4.004]
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.367, 95% CI [1.502 to 3.762]
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.894, 95% CI [1.835 to 4.609]
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.902, 95% CI 2-sided [1.829 to 4.657]
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.218, 95% CI [2.025 to 5.172]
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.153, 95% CI [1.375 to 3.394]
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.074, 95% CI [1.957 to 4.878]
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.050, 95% CI [1.310 to 3.228]
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.908, 95% CI [1.856 to 4.599]
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.113, 95% CI [1.349 to 3.332]
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.594, 95% CI [1.653 to 4.104]
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p = 0.005, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.891, 95% CI 2-sided [1.210 to 2.973]
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.314, 95% CI [2.108 to 5.265]
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.027, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.646, 95% CI [1.060 to 2.566]
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.347, 95% CI [1.507 to 3.683]
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p = 0.010, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.792, 95% CI 2-sided [1.153 to 2.799]
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.819, 95% CI [1.805 to 4.441]
Statistical Analysis 21: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.357, 95% CI [1.513 to 3.699]
Statistical Analysis 22: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.131, 95% CI [1.999 to 4.950]
Statistical Analysis 23: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 12; Test type: Superiority; p = 0.152, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.373, 95% CI [0.891 to 2.122]
Statistical Analysis 24: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.090, 95% CI [1.351 to 3.252]

10. Secondary Outcome: Number of Participants With Mean Percent Reduction of 100% in The Mean Frequency of Moderate, and Severe VMS From Baseline to Each Study Week Up to Week 12
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Baseline was the average number of moderate to severe VMS per 24 hours based on the non-missing values in the 10 days immediately prior to randomization. Participant has 100% reduction from baseline to each post baseline week for the frequency of moderate to severe VMS.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg
Number analyzed (Participants) | 167 | 166 | 167
Participants
  Week 1 | 1 | 1 | 3
  Week 2 | 3 | 8 | 4
  Week 3 | 5 | 4 | 11
  Week 4 | 3 | 10 | 17
  Week 5 | 3 | 12 | 11
  Week 6 | 9 | 12 | 17
  Week 7 | 9 | 13 | 18
  Week 8 | 10 | 17 | 22
  Week 9 | 9 | 14 | 18
  Week 10 | 11 | 17 | 25
  Week 11 | 9 | 15 | 28
  Week 12 | 9 | 15 | 25
Statistical Analysis 1: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 1; Test type: Superiority; p = 0.951, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 0.915, 95% CI [0.036 to 23.464]
Statistical Analysis 2: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 1; Test type: Superiority; p = 0.362, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.889, 95% CI 2-sided [0.364 to 58.864]
Statistical Analysis 3: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 2; Test type: Superiority; p = 0.138, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.775, 95% CI [0.785 to 12.870]
Statistical Analysis 4: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 2; Test type: Superiority; p = 0.704, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.342, 95% CI [0.291 to 6.914]
Statistical Analysis 5: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 3; Test type: Superiority; p = 0.741, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 0.798, 95% CI [0.194 to 3.079]
Statistical Analysis 6: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 3; Test type: Superiority; p = 0.134, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.292, 95% CI [0.809 to 7.443]
Statistical Analysis 7: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 4; Test type: Superiority; p = 0.062, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.474, 95% CI [1.039 to 15.712]
Statistical Analysis 8: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 4; Test type: Superiority; p = 0.004, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 6.184, 95% CI [2.025 to 26.875]
Statistical Analysis 9: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 5; Test type: Superiority; p = 0.028, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 4.217, 95% CI 2-sided [1.305 to 18.806]
Statistical Analysis 10: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 5; Test type: Superiority; p = 0.044, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.802, 95% CI [1.157 to 17.075]
Statistical Analysis 11: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 6; Test type: Superiority; p = 0.519, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.342, 95% CI [0.551 to 3.382]
Statistical Analysis 12: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 6; Test type: Superiority; p = 0.117, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.961, 95% CI [0.863 to 4.741]
Statistical Analysis 13: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 7; Test type: Superiority; p = 0.393, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.471, 95% CI [0.612 to 3.687]
Statistical Analysis 14: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 7; Test type: Superiority; p = 0.086, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.087, 95% CI [0.923 to 5.043]
Statistical Analysis 15: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 8; Test type: Superiority; p = 0.168, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.774, 95% CI [0.798 to 4.143]
Statistical Analysis 16: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 8; Test type: Superiority; p = 0.030, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.374, 95% CI [1.112 to 5.410]
Statistical Analysis 17: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 9; Test type: Superiority; p = 0.287, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.605, 95% CI 2-sided [0.681 to 3.971]
Statistical Analysis 18: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 9; Test type: Superiority; p = 0.080, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.108, 95% CI [0.936 to 5.076]
Statistical Analysis 19: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 10; Test type: Superiority; p = 0.247, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.599, 95% CI 2-sided [0.730 to 3.636]
Statistical Analysis 20: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 10; Test type: Superiority; p = 0.017, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.481, 95% CI [1.201 to 5.441]
Statistical Analysis 21: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 11; Test type: Superiority; p = 0.212, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.728, 95% CI [0.744 to 4.236]
Statistical Analysis 22: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 11; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.536, 95% CI [1.666 to 8.207]
Statistical Analysis 23: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 30 mg; Week 12; Test type: Superiority; p = 0.225, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.701, 95% CI [0.733 to 4.169]
Statistical Analysis 24: Comparison: Double-blind Period: Placebo vs Double-blind Period: Fezolinetant 45 mg; Week 12; Test type: Superiority; p = 0.006, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 3.049, 95% CI [1.420 to 7.125]

11. Secondary Outcome: Change From Baseline in The Mean Frequency of Moderate, and Severe VMS at Week 24
Description: as for outcome 1
Time Frame: Baseline and 24 weeks of fezolinetant exposure (week 36 for arms Placebo/Fezolinetant 30 mg and Placebo/Fezolinetant 45 mg)
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: VMS per day
Arm/Group | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 131 | 134 | 62 | 60
VMS per day | -7.86 (4.21) | -7.96 (4.53) | -9.01 (5.80) | -7.08 (5.40)

12. Secondary Outcome: Change From Baseline in The Mean Severity of Moderate, and Severe VMS at Week 24
Description: as for outcome 3
Time Frame: as for outcome 11
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 131 | 134 | 62 | 60
Score on a scale | -0.85 (0.88) | -0.90 (0.80) | -0.78 (0.85) | -0.95 (0.88)

13. Secondary Outcome: Number of Participants in Each Category of Patient's Global Impression of Change (PGIC) in VMS at Each Visit
Description: The PGI is comprised of 2 companion 1-item PRO measures analogous to the Clinical Global Impression (CGI) scales. These measures provide brief, stand-alone global assessments prior to and after initiating a study medication. Patient-perceived change from the initiation of treatment (PGI-C)-VMS is used to evaluate meaningful within-person changes over time in VMS. This measure provides patient-perceived change from the initiation of treatment.
  The PGI-C VMS asks: "Compared to the beginning of this study, how would you rate your HFs/night sweats now?" Subject ratings range from (1) much better to (7) much worse. Participant ratings range from 1=much better, 2= moderately better, 3= a little better, 4= no change, 5= a little worse, 6= moderately worse, 7= much worse.
Time Frame: Weeks 4, 12, 16, 20, 24, 28, 32, 36, 40, 44, 52 of fezolinetant exposure (weeks 16, 24, 28, 32, 36, 40, 44, 48 and 52 for arms Placebo/Fezolinetant 30 mg and Placebo/Fezolinetant 45 mg)
Population: FAS population with available data at specified time point.
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 151 | 155 | 159 | 67 | 69
Participants
  Week 4: Much better: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4: Much better | 25 | 61 | 68 |  | 2
  Week 4:Moderately better: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4:Moderately better | 23 | 21 | 32 |  | 0
  Week 4:A little better: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4:A little better | 46 | 42 | 42 |  | 1
  Week 4:No change: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4:No change | 43 | 29 | 16 |  | 0
  Week 4:A little worse: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4:A little worse | 6 | 2 | 0 |  | 0
  Week 4:Moderately worse: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4:Moderately worse | 6 | 0 | 0 |  | 0
  Week 4:Much worse: number analyzed (Participants) | 151 | 155 | 159 | 0 | 3
  Week 4:Much worse | 2 | 0 | 1 |  | 0
  Week 12: Much better: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: Much better | 35 | 68 | 71 | 40 | 30
  Week 12: Moderately better: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: Moderately better | 24 | 25 | 37 | 11 | 18
  Week 12: A little better: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: A little better | 36 | 29 | 32 | 11 | 10
  Week 12: No change: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: No change | 39 | 19 | 8 | 4 | 4
  Week 12: A little worse: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: A little worse | 6 | 1 | 1 | 1 | 4
  Week 12: Moderately worse: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: Moderately worse | 2 | 2 | 0 | 0 | 1
  Week 12: Much worse: number analyzed (Participants) | 151 | 145 | 149 | 67 | 69
  Week 12: Much worse | 2 | 1 | 0 | 0 | 2
  Week 16: Much better: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: Much better |  | 0 | 2 |  |
  Week 16: Moderately better: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: Moderately better |  | 0 | 0 |  |
  Week 16: A little better: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: A little better |  | 0 | 0 |  |
  Week 16: No change: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: No change |  | 0 | 0 |  |
  Week 16: A little worse: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: A little worse |  | 0 | 0 |  |
  Week 16: Moderately worse: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: Moderately worse |  | 0 | 0 |  |
  Week 16: Much worse: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
  Week 16: Much worse |  | 1 | 0 |  |
  Week 20: Much better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: Much better |  | 1 |  |  |
  Week 20: Moderately better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: Moderately better |  | 0 |  |  |
  Week 20: A little better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: A little better |  | 0 |  |  |
  Week 20: No change: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: No change |  | 1 |  |  |
  Week 20: A little worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: A little worse |  | 0 |  |  |
  Week 20: Moderately worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: Moderately worse |  | 0 |  |  |
  Week 20: Much worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 20: Much worse |  | 0 |  |  |
  Week 24: Much better: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: Much better |  | 68 | 76 | 0 |
  Week 24: Moderately better: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: Moderately better |  | 31 | 33 | 1 |
  Week 24: A little better: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: A little better |  | 22 | 22 | 0 |
  Week 24: No change: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: No change |  | 9 | 4 | 0 |
  Week 24: A little worse: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: A little worse |  | 1 | 3 | 0 |
  Week 24: Moderately worse: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: Moderately worse |  | 2 | 1 | 0 |
  Week 24: Much worse: number analyzed (Participants) | 0 | 134 | 139 | 1 | 0
  Week 24: Much worse |  | 1 | 0 | 0 |
  Week 28: Much better: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: Much better |  | 1 | 0 | 1 |
  Week 28: Moderately better: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: Moderately better |  | 0 | 0 | 0 |
  Week 28: A little better: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: A little better |  | 0 | 0 | 0 |
  Week 28: No change: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: No change |  | 0 | 0 | 0 |
  Week 28: A little worse: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: A little worse |  | 0 | 0 | 0 |
  Week 28: Moderately worse: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: Moderately worse |  | 0 | 0 | 0 |
  Week 28: Much worse: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 28: Much worse |  | 0 | 1 | 0 |
  Week 32: Much better: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Much better |  |  | 1 |  |
  Week 32: Moderately better: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Moderately better |  |  | 0 |  |
  Week 32: A little better: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: A little better |  |  | 0 |  |
  Week 32: No change: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: No change |  |  | 0 |  |
  Week 32: A little worse: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: A little worse |  |  | 0 |  |
  Week 32: Moderately worse: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Moderately worse |  |  | 0 |  |
  Week 32: Much worse: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Week 32: Much worse |  |  | 0 |  |
  Week 36: Much better: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: Much better |  | 0 |  |  |
  Week 36: Moderately better: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: Moderately better |  | 1 |  |  |
  Week 36: A little better: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: A little better |  | 0 |  |  |
  Week 36: No change: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: No change |  | 0 |  |  |
  Week 36: A little worse: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: A little worse |  | 0 |  |  |
  Week 36: Moderately worse: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: Moderately worse |  | 0 |  |  |
  Week 36: Much worse: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36: Much worse |  | 0 |  |  |
  Week 40: Much better: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: Much better |  |  |  | 33 | 31
  Week 40: Moderately better: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: Moderately better |  |  |  | 14 | 13
  Week 40: A little better: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: A little better |  |  |  | 5 | 8
  Week 40: No change: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: No change |  |  |  | 3 | 2
  Week 40: A little worse: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: A little worse |  |  |  | 0 | 0
  Week 40: Moderately worse: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: Moderately worse |  |  |  | 0 | 0
  Week 40: Much worse: number analyzed (Participants) | 0 | 0 | 0 | 55 | 54
  Week 40: Much worse |  |  |  | 0 | 0
  Week 44: Much better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: Much better |  | 2 |  |  |
  Week 44: Moderately better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: Moderately better |  | 0 |  |  |
  Week 44: A little better: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: A little better |  | 0 |  |  |
  Week 44: No change: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: No change |  | 0 |  |  |
  Week 44: A little worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: A little worse |  | 0 |  |  |
  Week 44: Moderately worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: Moderately worse |  | 0 |  |  |
  Week 44: Much worse: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Week 44: Much worse |  | 0 |  |  |
  Week 52: Much better: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: Much better |  | 60 | 77 |  |
  Week 52: Moderately better: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: Moderately better |  | 25 | 22 |  |
  Week 52: A little better: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: A little better |  | 14 | 13 |  |
  Week 52: No change: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: No change |  | 4 | 2 |  |
  Week 52: A little worse: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: A little worse |  | 1 | 0 |  |
  Week 52: Moderately worse: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: Moderately worse |  | 1 | 0 |  |
  Week 52: Much worse: number analyzed (Participants) | 0 | 107 | 116 | 0 | 0
  Week 52: Much worse |  | 2 | 2 |  |

14. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant administered a study drug, & which does not necessarily have to have a causal relationship with treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with use of a medicinal product (mp) whether or not considered related to the mp. An AE is considered "serious" if it results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, Results in congenital anomaly or birth defect, requires inpatient hospitalization or leads to prolongation of hospitalization, hospitalization for treatment/observation/examination caused by AE is to be considered as serious, discontinuation due to increases in liver enzymes, other medically important events. TEAE was defined as an AE observed from first dose date up to 21 days after last dose.
Time Frame: From first dose date up to 21 days after last dose (up to 55 weeks)
Population: Safety analysis set consisted of all randomized participants who took at least 1 dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
Number analyzed (Participants) | 167 | 166 | 167 | 76 | 75
Participants
  Treatment Emergent Adverse Events (TEAE) | 54 | 107 | 106 | 43 | 45
  Drug-related TEAE | 11 | 33 | 30 | 8 | 8
  Serious TEAE | 0 | 9 | 8 | 2 | 4
  Drug-related serious TEAE | 0 | 0 | 1 | 0 | 1
  TEAE leading to death | 0 | 0 | 0 | 0 | 1
  Drug-related TEAE leading to death | 0 | 0 | 0 | 0 | 0
  TEAE leading to withdrawal of treatment | 1 | 4 | 7 | 2 | 3
  Drug-related TEAE leading to withdrawal of treatment | 0 | 1 | 6 | 1 | 2
  Death | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose date up to 21 days after last dose (up to 55 weeks)
Arm/Group | Double-blind Period: Placebo | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/166 | 0/167 | 0/76 | 1/75
Serious Adverse Events (participants affected / at risk) | 0/167 | 9/166 | 8/167 | 2/76 | 4/75
Other Adverse Events (participants affected / at risk) | 6/167 | 20/166 | 34/167 | 10/76 | 12/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Placebo (N=167) | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg (N=166) | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg (N=167) | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg (N=76) | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg (N=75)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior tibial nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Placebo (N=167) | Double-blind Period: Fezolinetant 30 mg/Extension Period: Fezolinetant 30 mg (N=166) | Double-blind Period: Fezolinetant 45 mg/Extension Period: Fezolinetant 45 mg (N=167) | Double-blind Period: Placebo/Extension Period: Fezolinetant 30 mg (N=76) | Double-blind Period: Placebo/Extension Period: Fezolinetant 45 mg (N=75)
COVID-19 (Infections and infestations) | 1 (1) | 8 (8) | 15 (15) | 4 (4) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 5 (6)
Headache (Nervous system disorders) | 4 (4) | 8 (9) | 12 (14) | 1 (1) | 4 (5)
Hot flush (Vascular disorders) | 1 (1) | 3 (3) | 7 (7) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04003142/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04003142/SAP_001.pdf